CLINICAL TRIAL: NCT00006208
Title: A Randomized, Double-Blind, Equivalence Trial Comparing Emtricitabine to Stavudine Within a Triple Drug Combination Containing Didanosine Plus Efavirenz in Antiretroviral-Drug Naive HIV-1 Infected Patients
Brief Title: A Comparison of Emtricitabine and Stavudine Used With Didanosine Plus Efavirenz in HIV-Infected Patients Who Have Not Taken Anti-HIV Drugs
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Triangle Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 298C; FTC-301
Record Dates: First submitted 2000-09-11; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2006-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Didanosine; Drug Therapy, Combination; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Deoxycytidine; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Emtricitabine; Stavudine; Didanosine

INTERVENTIONS:
Drug: Efavirenz
Drug: Emtricitabine
Drug: Stavudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of emtricitabine and stavudine when given with didanosine plus efavirenz to HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old at the time of screening.
* Have plasma HIV-1 RNA loads (level of HIV in your blood) of 5,000 or more copies/ml at the time of screening.
* Have not used any anti-HIV therapy for more than 2 days.
* Have a negative pregnancy test within 22 days of starting study drugs.
* Can be reached by telephone.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.
* Use alcohol or illegal drugs that, in the opinion of the principal investigator, may interfere with the patient's ability to follow the dosing schedule and protocol evaluations.
* Are being treated for active tuberculosis.
* Are using astemizole, cisapride, midazolam, triazolam, ergot derivatives, St. John's wort, or drugs for a mental disorder.
* Have a history of a serious mental disorder.
* Are unwilling to use an effective barrier method of birth control during the study (for women who can get pregnant).
* Have a history of opportunistic infections and cancers (Mycobacterium avium complex, cytomegalovirus, toxoplasmic encephalitis or disseminated toxoplasmosis, cryptosporidiosis, Isospora belli, progressive multifocal leukoencephalopathy, visceral Kaposi's sarcoma, and lymphoma). Patients with past episode of pulmonary tuberculosis, Pneumocystis carinii pneumonia, or isolated cutaneous Kaposi's sarcoma are allowed. Medication for the prevention of PCP (TMP/SMX, nebulized pentamidine, and atovaquone) is allowed.
* Have peripheral neuropathy (a painful condition affecting the nervous system) or history of peripheral neuropathy.
* Cannot take medicine by mouth or have severe chronic diarrhea within 30 days before beginning the study.
* Cannot eat 1 or more meals a day because of chronic nausea, vomiting, or abdominal or esophageal discomfort.
* Have had a serious illness or injury within 30 days of screening. Treatment must have been completed for 14 days prior to study entry.
* Have a history of AIDS-defining opportunistic infection, except for tuberculosis or infection of the stomach or intestines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Locations (63):
- United States (51):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - East Bay AIDS Ctr, Berkeley, California
  - East Bay Clinical Trial Ctr, Concord, California
  - Mem Med Group Inc, Long Beach, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - Orange Coast Med Group, Newport Beach, California
  - St Lukes Medical Group, San Diego, California
  - Robert Smith Medical Group, San Diego, California
  - Saint Francis Mem Hosp / HIV Care, San Francisco, California
  - Davies Med Ctr, San Francisco, California
  - Beacon Clinic / Boulder Community Hosp, Boulder, Colorado
  - Univ of Colorado Health Ctr / Denver Gen Hosp, Denver, Colorado
  - Blick Med Associates, Stamford, Connecticut
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Physicans Home Service, Washington D.C., District of Columbia
  - Gary Richmond MD, Fort Lauderdale, Florida
  - South Miami Hosp, Miami, Florida
  - Wohlfeiler, Piperator & King, MD, PA, Miami Beach, Florida
  - Larry Bush, Palm Springs, Florida
  - Health Positive, Safety Harbor, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - Hillsborough County Health Department, Tampa, Florida
  - Infectious Disease Research Inst, Tampa, Florida
  - Ingenix Kern McNeill Decatur, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Harbin Clinic, Rome, Georgia
  - Northstar Med Clinic, Chicago, Illinois
  - Tulane Univ Med Ctr / Infectious Diseases Sect, New Orleans, Louisiana
  - Institute of Human Virology, Baltimore, Maryland
  - New England Med Ctr, Boston, Massachusetts
  - Fenway Community Health Ctr, Boston, Massachusetts
  - Abbott-Northwestern Hosp / Clinic 42, Minneapolis, Minnesota
  - South Jersey Infectious Diseases Inc, Somers Point, New Jersey
  - Erie County Med Ctr, Buffalo, New York
  - North Shore Univ Hosp / Div of Infectious Diseases, Manhasset, New York
  - Dr Lawrence Fontana, New York, New York
  - Liberty Medical / Cabrini Hospital / Dept of Infec Diseases, New York, New York
  - Howard Grossman, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Fanno Creek Clinic, Portland, Oregon
  - Paragon Clinical Research, Cranston, Rhode Island
  - Coastal Carolina Research Ctr, Mt. Pleasant, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - Nelson Tebedo Health Resource Ctr, Dallas, Texas
  - Amelia Ct Clinic, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Diversified Med Practices, PA, Houston, Texas
  - Walter Gaman, Irving, Texas
  - Swedish Med Ctr / Dr Peter Shalit, Seattle, Washington
- Argentina (5):
  - FUNCEI, Buenos Aires
  - Fundacion HUES, Buenos Aires
  - Hospital de Agudos JM Ramos Mejia, Buenos Aires
  - Hospital Muniz, Buenos Aires
  - Hospital Interzonal Gen de Agudos Oscar Alende, Mar del Plata
- Canada (4):
  - Viridae Clinical Sciences / University of British Columbia, Vancouver, British Columbia
  - McMaster Univ Med Centre, Hamilton, Ontario
  - Montreal Gen Hosp, Montreal, Quebec
  - Centre De Recherche En Infectiologie, Ste Foy, Quebec
- Fundacion Arriaran, Santiago, Chile
- Instituto Nacional de la Nutricion, Mexico City, Mexico
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico